CLINICAL TRIAL: NCT05867368
Title: Evaluating the Effect of Virtual Reality on the Upper-extremity Function of Children With Hemiplegic Cerebral Palsy Participating in Hand Arm Bimanual Training Camps
Brief Title: Hand-Arm Bimanual Intensive Therapy in Virtual Reality Versus Standard Hand-Arm Bimanual Intensive Therapy
Acronym: HABIT-VR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0154-22-EP
Record Dates: First submitted 2023-04-27; First posted 2023-05-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Hand Arm Bimanual Intensive Therapy; Virtual Reality

STUDY DESIGN:
Intervention Model Description: Participants are assigned based on which camp is being offered that summer. The investigators enroll on a first-come, first serve basis, until the camp is full.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard HABIT (Active Comparator): Children will receive hand arm bimanual intensive therapy the way it is typically delivered. Children will receive 40 hrs of one-on-one bimanual therapy, delivered as play. Activities will be self-selected, but all options will require both hands to succeed.
  Interventions: Behavioral: Standard HABIT
- HABIT-VR (Experimental): Children will receive hand arm bimanual intensive therapy, however, it will be through the use of custom virtual reality games. Children will receive 40 hrs of one-on-one bimanual therapy, delivered through the virtual reality games. Activities will be self-selected, but all games have a task constraint, requiring both hands to succeed.
  Interventions: Behavioral: HABIT-VR

INTERVENTIONS:
Behavioral: HABIT-VR — HABIT-VR is a suite of video games designed on the principals of HABIT treatments. The games are delivered in virtual reality, because these systems provide a way to track the movements of both hands and build software that requires both hands to succeed.
  Other Names: Hand arm bimanual intensive training in virtual reality
  Arms: HABIT-VR
Behavioral: Standard HABIT — HABIT is a camp where children play self-select activities that require both hands to succeed.
  Other Names: Hand arm bimanual intensive training
  Arms: Standard HABIT

SUMMARY:
The goal of this intervention study is- 1. To determine if a camp that solely uses VR software based on HABIT (HABIT-VR) still improves the motor planning and execution deficits in children with hemiplegic cerebral palsy (HCP) and 2. To determine if HABIT-VR improves bimanual coordination and affected hand function in children with HCP at least as well as a standard HABIT.

Children with motor planning and execution deficits will receive 40 hours of either HABIT-VR or standard HABIT (4 hours per day, 5days/week, for two consecutive weeks), during which the investigators will track their performance of the tasks and their movements through 3-D motion tracking of the VR system. Post-camp, again the investigators will assess upper-extremity motor function. Additionally the investigators will assess pre to post camp improvement in hand function and bimanual coordination using Assisting Hand Assessment (AHA), Manual Ability Classification System (MACS), and manual dexterity using Box and Block test and 9 Hole Peg test.

DETAILED DESCRIPTION:
The Physical or Occupational Therapist will first confirm the diagnosis of HCP and refer the child to PI after knowing parental willingness to participate in this investigation. The PI will screen the child for inclusion criteria, explain the purpose of study and procedures to the parents and obtain parental consent for their child's participation in the study.

The process of informed consent will take place in the Virtual Reality Laboratory in the Munroe-Meyer Institute (MMI), with all participants and their families being screened for Corona Virus Disease 2019 (COVID-19) at the entrance of MMI. All study personnel will be wearing the required protective equipment to go over the consent form. All procedures will be reviewed with the parents once again.

There will be two groups for this investigation, each group will participate in a single camp. One group/camp will be 100% HABIT-VR, the other group/camp will participate in a standard HABIT camp with zero VR. Subjects will be assigned to the 2022 camp on a first come first serve basis until the camp is full, the remaining subjects will participate in the 2023 camp.

After the parents sign the informed consent, the investigators will assess the hand function and bimanual coordination using the Box and Block test and 9 hole Peg test, both in the traditional environment and in a virtual environment, as a measure of manual dexterity. Additionally, the investigators will assess the hand function and bimanual coordination using Assisting Hand Assessment (AHA) for children with HCP. Video recordings of the AHA, BBT, and Nine Peg Hole Test sessions will be taken to validate test scores in post. Further, the participants will undergo Range of Motion, Grip Strength, and Functional Reach testing, all tests used in clinic and will be administered by our clinical research team members. The range of motion testing will quantify the degrees the patient can move their upper-extremity joints. The grip strength testing will have the participants squeeze a force measuring handle 3 times with each hand. The Functional Reach Test assesses a patient's stability by measuring the maximum distance an individual can reach forward while standing in a fixed position. The investigators will also collect baseline physiological responses during the pre-assessment. The child will wear an Empatica E4 device that records their skin temperature, their galvanic skin response, and their heart rate. These data will be used to compare to their physiological responses during the camp, to assess arousal levels and acceptability difference between the camps.

After the pre-assessment, the investigators will enroll children for 40 hrs HABIT-VR or standard HABIT, which will be conducted for 4 hrs/day, 5 days/week for two consecutive weeks. Both groups will occur as a summer camp for children with HCP. The children will be assigned in order of enrollment and the camps will be held serially. Two participating personnel per child will continuously monitor the child's activities. The parent will be required to stay at the research site each day during the 40 hrs camp session. The HABIT-VR camp will consists of various bimanual goal directed activities and functional training in a play context in VR, 4 hrs/day for 10 days. The children will play HABIT-VR games in 40 minute blocks with mandatory breaks every 30 minutes. The length of these breaks will be child driven, but will be at least 10 minutes, as suggested by the US Department of Business, Energy and Industrial Strategy. Additionally, the children will be taken to an indoor or outdoor playground for 30 minutes halfway through each day, to give them further extended breaks.In the standard HABIT camp, children will participate in self-selected activities that require both hands to succeed.

In both camps, the investigators will incorporate age-appropriate fine motor and manipulative gross motor activities that require the use of both hands. The investigators will select specific activities by considering the role of the involved limb in the activity (e.g. stabilizer, manipulator, active/passive assist). The investigators will grade the task demands to allow success, and the investigators will increase the task difficulty to increase the complexity of the task and allow variations in the practice. The investigators will record the task performance, and both positive reinforcement and knowledge of performance will be used to motivate performance and to reinforce target movements. The tasks delivered as VR games will record the individuals game score, along with the positions of their upper extremities and head while playing the game. The investigators will give instructions to the child before the start of each task in order to specify how each hand should be used during the activity and to avoid use of compensatory strategies (performing the task unimanually with the non-involved extremity). If a child attempts to use the non-involved hand inappropriately (e.g. using compensatory strategies as a substitution for involved hand use), the person who is monitoring a child will pause the task and a reminder of the task rules will be given to the child. Specific instructions will be given to the participating personnel to avoid urging the child to use his/her involved hand and avoid physically inhibiting use of the non-involved hand during an activity. The investigators will engage children in two types of structured practice during the HABIT-VR: whole task and part task practice. During performance of whole task practice, activities will be performed continuously for at least 15 to 20 minutes but no longer than 1 hour. Targeted movements and spatial and temporal movement coordination will be practiced within the context of completing a task (e.g. playing a board game). Part task practice will involve practicing a targeted movement exclusive of other movements. Specifically, symmetrical bimanual movements will be often used to elicit a targeted movement (e.g. putting game pieces away simultaneously with each hand) because of the simplicity of control. One participating person will record the frequency of successful task completion (the number of times the child succeeded in 30s) while the other person will engage the child in the activities. Participating person will increase the task difficulty by increasing speed and accuracy of the task. Additionally, they will incorporate tasks that require more skilled use of the involved hand and arm (e.g. moving from activities in which the involved limb acted as a stabilizer to activities that required manipulative skills). Participating personal monitoring each child will emphasize on completing each movement with the involved upper extremity in the same way as the non-dominant hand of a typically developing child (i.e. as a stabilizer or manipulator). Practice will be structured to promote increased intensity: the involved hand will not be merely used to assist in every activity. Children will also wear an Empatica E4 physiological recording device during the camp, to record their physiological responses to the different camps. The investigators will conduct make up sessions if a child is not able to participate any day/days during the camp for 4 hrs.

At the end of each day, the children will be surveyed to assess their acceptability of the camp environments. These surveys will be 7 point likert scales that ask them questions about how they enjoyed the games and their fatigue levels. These data will be used in combination with the physiological recordings to validate if their arousal responses align with their survey responses.

The investigators will once again perform AHA, Box and Block test, and 9 Hole Peg test to assess bimanual function and manual dexterity respectively after both camps. Again, video recordings of the AHA, BBT, and 9HPT sessions will be taken to validate test scores in post. Additionally, the investigators will assess kinematics of reaching to evaluate changes in movement velocities, looking at both the effect of the camp and the difference between the groups. This study consists of a total of 12 research visits. Pre-intervention, the first research visit will consists of the assessment of kinematics of the arm and hand, the testing of hand function using Box and Block test, 9 hole peg test, AHA test. This research visit will be of a total 2 hrs. The pre-assessment visits will be done within one week prior to the start of both camps. The camps will consists of 4 hrs daily sessions for 5 days/week, for 2 consecutive weeks. Post-camp, children will have one assessment session. During the post-assessment research visit, the investigators will assess the kinematics, Box and Block test, Purdue Pegboard test, and the AHA. The post-camp sessions will consists of 2 hrs. Physiological recordings with an Empatica E4 will occur during the post-assessments. The parent(s) will be required to accompany the child during the pre- and post-assessment sessions.

After the conclusion of the data analysis, the video recordings of the AHA, 9HPT, and BBT will be deleted.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as HCP.
* Children with HCP having Manual Ability Classification System Score (MACS) between I-IV.
* Parents able to give consent for the assessment and willing to adhere to the assessment and HABIT protocol.

Exclusion Criteria:

* Children with any other neurological conditions such as diplegic or tetraplegic cerebral palsy CP, birth injuries such as erbs palsy, brachial plexus lesion or peripheral nerve injuries, spina bifida at the upper thoracic level, leading to inability to move the upper extremity.
* Children with known visual impairments such as blindness.
* Children with any obvious musculoskeletal deformity, which will affect the ability to handle objects.
* Children with musculoskeletal problems such as torticollis, which will affect visual gaze and visual tracking of an object.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Assisting Hand Assessment Score | Approximately 1 week before the camp
  The Assisting Hand Assessment (AHA)measure and describe how effectively individuals with a hand/arm impairment use their two hands together to perform bimanual tasks.
  The scale range from 22 points, meaning that the hand is not used at all, to 88 points meaning that the hand is used effectively, like a normal non-dominant hand. The score reflects the child's ability to use the affected hand in bimanual performance. Higher scores are better.
Assisting Hand Assessment Score | Approximately 1 week after the camp
  The Assisting Hand Assessment (AHA)measure and describe how effectively individuals with a hand/arm impairment use their two hands together to perform bimanual tasks. The scale range from 22 points, meaning that the hand is not used at all, to 88 points meaning that the hand is used effectively, like a normal non-dominant hand. The score reflects the child's ability to use the affected hand in bimanual performance. Higher scores ar better.
Box and Blocks Score | Approximately 1 week before the camp
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. Children move blocks from one box to another in a minute. The minimum score is zero and there is no maximum score, as the blocks get reset if the child runs out. Higher scores are better.
Box and Blocks Score | Approximately 1 week after the camp
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. Children move blocks from one box to another in a minute. The minimum score is zero and there is no maximum score, as the blocks get reset if the child runs out. Higher scores are better.
9-Hole Peg Test Score | Approximately 1 week before the camp
  The Nine-Hole Peg Test (9-HPT) is a standardized, quantitative assessment used to measure finger dexterity. Children pick up pegs and try to place them in holes on a game board. The minimum score is zero and there is no maximum score, as it is a rate per second of how fast the child places the pegs. Lower scores are better.
9-Hole Peg Test Score | Approximately 1 week after the camp
  The Nine-Hole Peg Test (9-HPT) is a standardized, quantitative assessment used to measure finger dexterity. Children pick up pegs and try to place them in holes on a game board. The minimum score is zero and there is no maximum score, as it is a rate per second of how fast the child places the pegs. Lower scores are better.

SECONDARY OUTCOMES:
Heart Rate | Approximately 1 week before the camp for 5 minutes
  The investigators are collecting heart rate using an Empatica E4 during the camps. Heart rate is the number of heartbeats per minute. The typical heart rate for the age range included in this study is as follows:
  Children 6 years old: 75 to 115 beats per minute Children 7 to 9 years old: 70 to 110 beats per minute Children 10 years and older: 60 to 100 beats per minute
  The sensor measuring heart rate will use infrared light to measure the speed of blood as it moves through the arteries. This is non-invasive.
Heart Rate | During the camp up to 40 hours
  The investigators are collecting heart rate using an Empatica E4 during the camps. Heart rate is the number of heartbeats per minute. The typical heart rate for the age range included in this study is as follows:
  Children 6 years old: 75 to 115 beats per minute Children 7 to 9 years old: 70 to 110 beats per minute Children 10 years and older: 60 to 100 beats per minute
  The sensor measuring heart rate will use infrared light to measure the speed of blood as it moves through the arteries. This is non-invasive.
Heart Rate | Approximately 1 week after the camp for 5 minutes
  The investigators are collecting heart rate using an Empatica E4 during the camps. Heart rate is the number of heartbeats per minute. The typical heart rate for the age range included in this study is as follows:
  Children 6 years old: 75 to 115 beats per minute Children 7 to 9 years old: 70 to 110 beats per minute Children 10 years and older: 60 to 100 beats per minute
  The sensor measuring heart rate will use infrared light to measure the speed of blood as it moves through the arteries. This is non-invasive.
Galvanic Skin Response | Approximately 1 week before the camp for 5 minutes
  The investigators are collecting galvanic skin responses using an Empatica E4 during the camps. Two electrodes on the watch will press against the skin on the wrist. A low level, and imperceivable signal will be sent between these electrodes to measure the conductivity of the skin.
  Galvanic Skin Response (GSR) is a physiological measure that has been used in research for over a century. GSR measures the electrical conductance of the skin, which changes in response to emotional arousal and other psychological processes. This non-invasive method has proven to be a useful tool in understanding the mechanisms behind emotional responses and assessing psychological states.
Galvanic Skin Response | During the camp up to 40 hours
  The investigators are collecting galvanic skin responses using an Empatica E4 during the camps. Two electrodes on the watch will press against the skin on the wrist. A low level, and imperceivable signal will be sent between these electrodes to measure the conductivity of the skin.
  Galvanic Skin Response (GSR) is a physiological measure that has been used in research for over a century. GSR measures the electrical conductance of the skin, which changes in response to emotional arousal and other psychological processes. This non-invasive method has proven to be a useful tool in understanding the mechanisms behind emotional responses and assessing psychological states.
Galvanic Skin Response | Approximately 1 week after the camp for 5 minutes
  The investigators are collecting galvanic skin responses using an Empatica E4 during the camps. Two electrodes on the watch will press against the skin on the wrist. A low level, and imperceivable signal will be sent between these electrodes to measure the conductivity of the skin.
  Galvanic Skin Response (GSR) is a physiological measure that has been used in research for over a century. GSR measures the electrical conductance of the skin, which changes in response to emotional arousal and other psychological processes. This non-invasive method has proven to be a useful tool in understanding the mechanisms behind emotional responses and assessing psychological states.
Skin Temperature | Approximately 1 week before the camp for 5 minutes
  The investigators are collecting skin temperature using an Empatica E4 during the camps. This will be measured using a sensor that utilizes infrared light. The normal level for adults is between 92.3 and 98.4 Fahrenheit or 33-37 Celsius for peripheral skin temperature. This gives a measure of vasodilation, which can be used to measure stress or excitement.
Skin Temperature | During the camp up to 40 hours
  The investigators are collecting skin temperature using an Empatica E4 during the camps. This will be measured using a sensor that utilizes infrared light. The normal level for adults is between 92.3 and 98.4 Fahrenheit or 33-37 Celsius for peripheral skin temperature. This gives a measure of vasodilation, which can be used to measure stress or excitement.
Skin Temperature | Approximately 1 week after the camp for 5 minutes
  The investigators are collecting skin temperature using an Empatica E4 during the camps. This will be measured using a sensor that utilizes infrared light. The normal level for adults is between 92.3 and 98.4 Fahrenheit or 33-37 Celsius for peripheral skin temperature. This gives a measure of vasodilation, which can be used to measure stress or excitement.

CONTACTS AND LOCATIONS:
Overall Officials: James E Gehringer, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Munroe-Meyer Institute, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical outcome measures and physiological responses will be made available after completion of the study.
Supporting Information: CSR
Time Frame: De-identified data will be released after conclusion of data collections (planned for mid 2024), conclusion of data analysis (planned for end of 2024), and submission of publication (planned for end of 2024/early 2025)
Access Criteria: Data will be made available upon reasonable request.
URL: https://www.unmc.edu/mmi/research/virtual-reality-lab.html

REFERENCES:
- [Background] Gehringer JE, Fortin E, Surkar SM, Hao J, Pleiss M, Jensen-Willett S. Hand-Arm Bimanual Intensive Training in Virtual Reality: A Feasibility Study. Pediatr Phys Ther. 2023 Jan 1;35(1):85-91. doi: 10.1097/PEP.0000000000000975. Epub 2022 Dec 2. PMID 36459077